CLINICAL TRIAL: NCT02645383
Title: An Observational Prospective Study of Comparing Pain Responses With Pattern Laser Platform and Conventional Laser System During the Panretinal Photocoagulation in Proliferative Diabetic Retinopathy
Brief Title: PASCAL Laser Platform Produces Less Pain Responses Compared To Conventional Laser System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocatepe University (Other)
Responsible Party: Principal Investigator, Umit Ubeyt INAN, Professor Doctor, Kocatepe University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0112S299
Record Dates: First submitted 2015-12-19; First posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Diabetic Retinopathy
Keywords: Pattern scan laser; Proliferative diabetic retinopathy; Pain
MeSH Terms: conditions — Diabetic Retinopathy; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PASCAL group (Active Comparator): Patients undergone PASCAL laser photocoagulation
  Interventions: Device: PASCAL laser
- Conventional group (Active Comparator): Patients undergone conventional laser photocoagulation
  Interventions: Device: Conventional laser

INTERVENTIONS:
Device: PASCAL laser — A novel semi-automatic and multi-shot photocoagulator called as PASCAL (Pattern scan laser, Opti-Medica Corp., Santa Clara, California, USA) was introduced with a reduction in pulse duration of each laser spot from typical 100 ms down to 10-30 millisecond. Compared with the conventional laser, shorter pulses have been shown to significantly reduce the risk of damage to the adjacent retinal tissues. One eye was treated with PASCAL laser, the other was treated with conventional laser with 30 minutes resting intervals. To avoid a bias about orientation or becoming accustomed to laser procedure, PASCAL laser was performed in the first eyes in half of the patients (14 patients) randomly.
  Arms: PASCAL group
Device: Conventional laser — Maintaining of good glycemic regulation and performing panretinal laser photocoagulation (PRP) with conventional laser device (ELLEX Integre, Adailade, Australia) when it is indicated are evidence based effective methods for proliferative diabetic retinopathy.One eye was treated with conventional laser, the other was treated with PASCAL laser with 30 minutes resting intervals. To avoid a bias about orientation or becoming accustomed to laser procedure, conventional laser was performed in the first eyes in half of the patients (14 patients) randomly.
  Arms: Conventional group

SUMMARY:
The aim of this study is to compare the severity of expressed pain scores in patients with PDR who underwent either PASCAL or conventional laser and to assess the association between patient characteristics and severity of pain.

DETAILED DESCRIPTION:
Proliferative diabetic retinopathy (PDR) is a severe complication of diabetes mellitus characterized by new vessel formation in the retina and optic disc. Tight glycemic control and laser treatment in the early phases of the disease may slow the progression of PDR. Panretinal photocoagulation (PRP) is a laser-based treatment modality that destroys the outer retina layers and thereby improves the oxygen supply of the inner retina. During the following years, sequential improvements took place, including introduction of yellow, green, and diode lasers with various advantages of each wavelength.

In 2006, a novel semi-automatic and multi-shot photocoagulator called as PASCAL (Pattern scan laser, Opti-Medica Corp., Santa Clara, California, USA) was introduced with a reduction in pulse duration of each laser spot from typical 100 ms down to 10-30 millisecond. Compared with the conventional laser, shorter pulses have been shown to significantly reduce the risk of damage to the adjacent retinal tissues.

Almost all patients experience pain during PRP. While some patients may tolerate the pain, the majority does not. One study reported that 64.1% of patients did not complete treatment due to pain and therefore had an increased risk of vision loss. To improve patient compliance, several anesthetic and analgesic techniques such as peribulbar anesthesia, oral anesthesia and topical eye drops have been used. The patient comfort, and thus compliance, may be improved by using the shorter exposure burns, avoiding red or infrared wavelengths with deeper penetration, and by decreasing overall treatment time.

The aim of the current study was to compare the severity of expressed pain scores in patients with PDR who underwent either PASCAL or conventional laser.

As a method of this study, both eyes were treated within the same session and while one eye was treated with PASCAL laser, the other was treated with conventional laser (ELLEX Integre, Adailade, Australia) with 30 minutes resting intervals. To avoid a bias about orientation or becoming accustomed to laser procedure, PASCAL laser was performed in the first eyes in half of the patients (14 patients) and conventional laser was performed in the first eyes in the other half of the patients randomly. While the spot size used to obtain a white-grayish spot on the retina was 200-400 µm in both PASCAL and conventional laser, the pulse duration was 100 ms with conventional laser and 30ms with PASCAL laser. In order to accurately and reliable compare the grade of pain between each procedures, the retinal areas and total number of spots were standardized. Similar numbers of laser spots were created by two laser systems in same retinal quadrants in both eyes. Ten minutes after the procedure ended the severity of pain was assessed using a verbal rating scale and a visual analog scale (VAS). In the verbal scale the patient rates the pain on a Likert scale verbally, e.g. "none", "mild pain", "moderate pain", "severe pain" or "very severe pain" in five grading system (0-4) and in the VAS they specify the severity of pain by indicating a position along a continuous line from 0 to 10. Using these scores, relationship between severity of pain and patient characteristics including history of prior PRP treatment (experience), gender and duration of diabetes mellitus were assessed. Patients were assigned either in the experienced or non-experienced groups depending on history of prior PRP.

ELIGIBILITY:
Inclusion Criteria:

* Patients (>18 years) with type 1 or 2 diabetes and bilateral high-risk proliferative diabetic retinopathy (PDR)

Exclusion Criteria:

* Patients with a history of focal/grid photocoagulation, a history of orbital trauma, orbital infection or surgery, those with corneal or lens opacities, those with vitreous hemorrhage and non-compliant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Verbal Score for pain | 3 months
  Verbal Score for pain was measured as units on the scale 10 minutes after the completion the laser procedure.
Visual analog score for pain | 3 months
  Visual Analog Score for pain was measured as units on the scale 10 minutes after the completion the laser procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Umit U Inan, M.D, Principal Investigator — Kocatepe University Medical School Department of Ophthalmology

REFERENCES:
- [Result] Aiello LP, Gardner TW, King GL, Blankenship G, Cavallerano JD, Ferris FL 3rd, Klein R. Diabetic retinopathy. Diabetes Care. 1998 Jan;21(1):143-56. doi: 10.2337/diacare.21.1.143. No abstract available. PMID 9538986
- [Result] Feman SS, Chen J, Burroughs TE. Change in diabetic panretinal photocoagulation incidence. Ophthalmic Surg Lasers Imaging. 2012 Jul 1;43(4):270-4. doi: 10.3928/15428877-20120618-02. PMID 22788579
- [Result] Jain A, Blumenkranz MS, Paulus Y, Wiltberger MW, Andersen DE, Huie P, Palanker D. Effect of pulse duration on size and character of the lesion in retinal photocoagulation. Arch Ophthalmol. 2008 Jan;126(1):78-85. doi: 10.1001/archophthalmol.2007.29. PMID 18195222
- [Result] Blumenkranz MS, Yellachich D, Andersen DE, Wiltberger MW, Mordaunt D, Marcellino GR, Palanker D. Semiautomated patterned scanning laser for retinal photocoagulation. Retina. 2006 Mar;26(3):370-6. doi: 10.1097/00006982-200603000-00024. No abstract available. PMID 16508446
- [Result] Zakrzewski PA, O'Donnell HL, Lam WC. Oral versus topical diclofenac for pain prevention during panretinal photocoagulation. Ophthalmology. 2009 Jun;116(6):1168-74. doi: 10.1016/j.ophtha.2009.01.022. Epub 2009 Apr 19. PMID 19376588
- [Result] Wu WC, Hsu KH, Chen TL, Hwang YS, Lin KK, Li LM, Shih CP, Lai CC. Interventions for relieving pain associated with panretinal photocoagulation: a prospective randomized trial. Eye (Lond). 2006 Jun;20(6):712-9. doi: 10.1038/sj.eye.6701989. Epub 2005 Jul 8. PMID 16021194
- [Result] Alvarez-Verduzco O, Garcia-Aguirre G, Lopez-Ramos Mde L, Vera-Rodriguez S, Guerrero-Naranjo JL, Morales-Canton V. Reduction of fluence to decrease pain during panretinal photocoagulation in diabetic patients. Ophthalmic Surg Lasers Imaging. 2010 Jul-Aug;41(4):432-6. doi: 10.3928/15428877-20100525-02. Epub 2010 May 28. PMID 20608612
- [Result] Schuele G, Rumohr M, Huettmann G, Brinkmann R. RPE damage thresholds and mechanisms for laser exposure in the microsecond-to-millisecond time regimen. Invest Ophthalmol Vis Sci. 2005 Feb;46(2):714-9. doi: 10.1167/iovs.04-0136. PMID 15671304
- [Result] Mainster MA. Decreasing retinal photocoagulation damage: principles and techniques. Semin Ophthalmol. 1999 Dec;14(4):200-9. doi: 10.3109/08820539909069538. PMID 10758220
- [Result] Al-Hussainy S, Dodson PM, Gibson JM. Pain response and follow-up of patients undergoing panretinal laser photocoagulation with reduced exposure times. Eye (Lond). 2008 Jan;22(1):96-9. doi: 10.1038/sj.eye.6703026. Epub 2007 Nov 23. PMID 18034195
- [Result] Nagpal M, Marlecha S, Nagpal K. Comparison of laser photocoagulation for diabetic retinopathy using 532-nm standard laser versus multispot pattern scan laser. Retina. 2010 Mar;30(3):452-8. doi: 10.1097/IAE.0b013e3181c70127. PMID 20216293
- [Result] Muqit MM, Marcellino GR, Gray JC, McLauchlan R, Henson DB, Young LB, Patton N, Charles SJ, Turner GS, Stanga PE. Pain responses of Pascal 20 ms multi-spot and 100 ms single-spot panretinal photocoagulation: Manchester Pascal Study, MAPASS report 2. Br J Ophthalmol. 2010 Nov;94(11):1493-8. doi: 10.1136/bjo.2009.176677. Epub 2010 Jun 16. PMID 20558423